# **SYNOPSIS**

# **Study Coronary bifurcation lesions 0-0-1**

# **Title and Study Name**

Coronary bifurcation lesions 0-0-1

# **Study Description**

Observational, non-interventional, retrospective, multicentric, non-randomized registry focused on the treatment of bifurcation lesions type 0-0-1 in current practice.

#### **Study Purpose**

To seek a clinical correlation with the angiographic analysis results of different angioplasty techniques used for the treatment of type 0-0-1 bifurcation lesions.

# **Device in Study**

N/A

#### **Number of Patients**

300 patients

# **Number of Centers**

- 1. Hôpital Jacques Cartier, Ramsay Général de Santé, Massy, France
- 2. Clinique Pasteur, Toulouse, France
- 3. Maasstad Hospital, Rotterdam, Netherlands

#### **Study Duration**

Follow-up (at 1 year and at the last possible follow-up) of patients who underwent angioplasty for a type 0-0-1 bifurcation lesion between 2016 and 2022.

#### Follow-up Methods

Patients will be contacted by phone to assess their clinical status, complications and events, examinations, and procedures that occurred after the angioplasty.

#### **Inclusion Criteria**

Any patient:

- Male or female aged 18 years and older
- Who underwent angioplasty for a type 0-0-1 coronary bifurcation lesion between 2016 and 2022

#### **Exclusion Criteria**

Any patient:

- Opposing the collection and processing of necessary data and refusing additional telephone follow-up

# **SYNOPSIS**

### **Primary Objective**

Combined criterion (Major Adverse Cardiac Event) including all-cause mortality, myocardial infarction, and target vessel revascularization [TVR].

# **Secondary Objectives**

- Separate analysis of mortality, myocardial infarction, and target vessel revascularization
- Analysis of a clinical evaluation score before and after angioplasty

# **Clinical Report**

The clinical report of the study will be based on the results at 12 months.

# **Sponsor**

Dr. Francesca Sanguineti Institut Cardiovasculaire Paris Sud Hôpital Privé Jacques Cartier 6 avenue du Noyer Lambert 91300 Massy, France